CLINICAL TRIAL: NCT01601483
Title: Phase II/III Study of the Efficacy and Safety of Macuclear MC-1101 1% TID in the Treatment of Nonexudative Age-Related Macular Degeneration
Brief Title: Efficacy and Safety Study of MC-1101 1% TID in the Treatment of Nonexudative Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unmasked without Sponsor's prior knowledge or authorization by the PI.
Sponsor: MacuCLEAR, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MacuCLEAR MC-1101-001
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Nonexudative Age Related Macular Degeneration
Keywords: AMD; Dry AMD; Nonexudative AMD; MC-1101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MC-1101 1% Ophthalmic Solution (Experimental)
  Interventions: Drug: MC-1101
- Vehicle control (Placebo Comparator)
  Interventions: Drug: MC-1101 Vehicle

INTERVENTIONS:
Drug: MC-1101 — 1% Ophthalmic Solution TID
  Arms: MC-1101 1% Ophthalmic Solution
Drug: MC-1101 Vehicle — Ophthalmic solution, TID
  Arms: Vehicle control

SUMMARY:
This is a Phase II/III vehicle controlled, double masked, single center study. A single eye of 60 individuals with mild to moderate nonexudative Age-Related Macular Degeneration (AMD) will be randomly assigned to receive either topical 1% MC-1101 or a vehicle control over 2 years. The study design will assess the efficacy, safety, and tolerability of MC-1101 for these patients.

An analysis of the primary and secondary endpoints will be conducted when all subjects have completed 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age ≥ 50 years and ≤ 85 years;
* Females must be at least 1 year postmenopausal (after last menstrual period) or sterilized;
* Better than 20/80 ETDRS best corrected visual acuity;
* Mild to moderate nonexudative AMD (AMD steps 3 through 8 on Age-Related Eye Disease Study (AREDS) Report No. 17 grading scale);
* Willing to sign informed consent, comply with study protocol requirements, and undergo up to 2.5 hours of testing at each visit;

Exclusion Criteria:

* Past or current exudative AMD or any geographic atrophy (on fundus autofluorescence) in study eye;
* Past or current other retinal or choroidal vasculopathy in study eye (e.g. pigment epithelial detachment, polypoidal choroidal vasculopathy, central serous retinopathy, retinal vein occlusion, sickle cell retinopathy);
* Uncontrolled hypertension (≥ 150 systolic or ≥95 diastolic);
* Diabetes mellitus;
* Glaucoma;
* Lens opacity ≥ grade 3 ARLNS on standard photographs;
* Unable to complete biophysical testing;
* Unable to give informed consent;
* Dilated pupil diameter less than 6 millimeters;
* Subjects with a history of a hypersensitivity reaction to the study drug or to any agent used in the components of the study assessment;
* Use of topical ocular medications (other than artificial tear products);
* Anticipated extra- or intraocular intervention during the study period;
* High myopia (refractive error spherical equivalent ≥ -6 diopters);
* Optic neuropathy;
* Neurological conditions that can impair vision (e.g. Parkinson's disease, multiple sclerosis, Alzheimer's disease);
* Liver disease (e.g. cirrhosis, hepatitis);
* History of GI surgery (e.g. bariatric surgery);
* Unwilling or unable to take an AREDS formula vitamin (without beta-carotene/vitamin A);
* Current or past use of chloroquine, hydroxychloroquine, chlorpromazine, thioridazine, quinine sulfate, clofazimine, cisplatin, carmustine (BCNU), or deferoxamine;
* Tobacco smoking (currently or within past 5 years);
* Contact lens wearers (not prepared to discontinue lens use);
* Ophthalmic surgery of any kind within 3 months prior to screening visit;
* Participation in any interventional clinical study requiring IRB approval within 3 months of enrollment;
* Currently being treated for cancer or any disease likely to adversely affect participation in a 2 year study;
* Known to have AIDS/HIV

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual Function | 12 months
  Primary efficacy assessment will be a comparison between groups of the change in visual function at 12 months with additional analyses at 18 and 24 months.

SECONDARY OUTCOMES:
Safety and Tolerability (incidence and severity of adverse events, ocular irritability, ocular hyperemia) | 24 months
  Evaluate the safety and tolerability (incidence and severity of adverse events, ocular irritability,and ocular hyperemia) of MC-1101 compared to vehicle control at each study visit following treatment for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Grant M Comer, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States